CLINICAL TRIAL: NCT01561547
Title: Maternal Analgesia for Procedural Pain in Preterm Neonates: Does It Remain Efficacious?
Brief Title: Trial of Repeated Analgesia With Kangaroo Care
Acronym: TRAKC
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: IWK Health Centre (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Nova Scotia Health Research Foundation (Other Government); Mayday Fund (Other)
Responsible Party: Principal Investigator, Celeste Johnston, Principal Investigator, IWK Health Centre
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TRAKC; CIHR-NSHRF-Mayday RPP 2446 (Other: CIHR-NSHRF-Mayday Fund RPP 244640)
Record Dates: First submitted 2012-03-08; First posted 2012-03-23 (Estimated); Last update posted 2016-09-20 (Estimated); Status verified 2016-09

CONDITIONS: Pain; Development
Keywords: pain; preterm neonate; sucrose; kangaroo mother care
MeSH Terms: conditions — Pain | interventions — Kangaroo-Mother Care Method; Sucrose

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Kangaroo Mother Care (Experimental): Infant is held in skin-to-skin contact with mother at least 15 minutes prior to painful procedure, remains in that position throughout the procedure and after the procedure at least until heart rate returns to baseline. Infant is given sterile water by mouth. This is for every heel lance and venipuncture, and if possible for tape removal.
  Interventions: Behavioral: Kangaroo Mother Care
- Sucrose (Active Comparator): Two minutes before the painful procedure and at the moment of the procedure, the infant will be given 24% sucrose by mouth. The volume is determined by body weight and is not important in terms of efficacy, it is the percentage of sweetness that is important.
  Interventions: Dietary Supplement: Sucrose
- Combination Kangaroo Mother Care and Sucrose (Experimental): Infant is held in skin-to-skin contact with mother at least 15 minutes prior to painful procedure, remains in that position throughout the procedure and after the procedure at least until heart rate returns to baseline. Infant is given sucrose water by mouth. This is for every heel lance and venipuncture, and if possible for tape removal.
  Interventions: Behavioral: Kangaroo Mother Care; Dietary Supplement: Sucrose

INTERVENTIONS:
Behavioral: Kangaroo Mother Care — Infant wearing only diaper is held in skin-to-skin contact with mother with flannel blanket around both mother and infant. removal.
  Arms: Combination Kangaroo Mother Care and Sucrose; Kangaroo Mother Care
Dietary Supplement: Sucrose — 24% sucrose in volumes between .05 to 2 ml depending on weight of the infant, is inserted by dropper into the infants mouth two minutes before and/or during the painful procedure with up to 3 doses.
  Arms: Combination Kangaroo Mother Care and Sucrose; Sucrose

SUMMARY:
Mothers can provide pain relief to their newborns, even in the context of intensive neonatal care. There is a recent accumulation of data, being analyzed by ourselves in a Cochrane review, that mothers holding their infants in a bare-chested skin-to-skin position, known as Kangaroo Mother Care (KMC), is effective in diminishing pain response during a single painful procedure. While evidence is compelling, leading to recommendations for its use, to date there is not a single study on the repeated efficacy to reduce pain. Current guidelines recommend sweet taste for minor painful procedures. Although there is some controversy about its continued use in this population based on one study with negative neurodevelopmental outcomes as well as its potential interaction with dopaminergic development, oral sucrose (sweet taste) remains efficacious in decreasing pain response over several weeks. The combination of KMC and sucrose is marginally more potent, but again, long term use remains unstudied.

AIMS. To test the repeated efficacy in diminishing pain from heel lance of KMC compared to usual care (sucrose), and of KMC in combination with sucrose by examining each condition at least three times during NICU stay. A secondary aim is to compare these interventions on neurodevelopment at discharge from the NICU.

ELIGIBILITY:
Inclusion Criteria:

* less than 36.0 weeks gestational age
* mother is generally available to provide kangaroo mother care

Exclusion Criteria:

* narcotic analgesics
* surgery in past 48 hrs
* major congenital anomalies

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 242 (Actual)
Dates: Start 2012-06; Primary Completion 2016-03 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Premature Infant Pain Profile (PIPP) | At the moment of painful procedure
  The PIPP is a composite measure of procedural pain and is based on changes from baseline in maximum heart rate and minimum oxygen saturation, and the duration of three facial actions. Data are analyzed in 30 second blocks from the moment the painful procedure begins. Time to return to baseline will also be noted. Scoring is done by assessors blind to the purpose of the study and group assignment.

SECONDARY OUTCOMES:
Neurobehavioral Assessment of Preterm Infants (NAPI) | 32, 36 and 40 weeks gestational age
  Two scales of the NAPI will be scored by person blinded to the intervention. These are 1) Motor Development and Vigour and 2) Alertness and Orientation

CONTACTS AND LOCATIONS:
Overall Officials: Celeste Johnston, RN, DEd, Principal Investigator — IWK Health Centre; Marsha Campbell-Yeo, RN, NNP, PhD, Study Director — IWK Health Centre
Locations (1):
- IWKHealthC, Halifax, Nova Scotia, Canada

IPD SHARING:
Plan to Share IPD: No
Aggregate data will be available but no individual data will be provided.

REFERENCES:
- [Background] Johnston CC, Campbell-Yeo M, Filion F. Paternal vs maternal kangaroo care for procedural pain in preterm neonates: a randomized crossover trial. Arch Pediatr Adolesc Med. 2011 Sep;165(9):792-6. doi: 10.1001/archpediatrics.2011.130. PMID 21893645
- [Background] Johnston CC, Filion F, Campbell-Yeo M, Goulet C, Bell L, McNaughton K, Byron J, Aita M, Finley GA, Walker CD. Kangaroo mother care diminishes pain from heel lance in very preterm neonates: a crossover trial. BMC Pediatr. 2008 Apr 24;8:13. doi: 10.1186/1471-2431-8-13. PMID 18435837
- [Background] Johnston CC, Stevens B, Pinelli J, Gibbins S, Filion F, Jack A, Steele S, Boyer K, Veilleux A. Kangaroo care is effective in diminishing pain response in preterm neonates. Arch Pediatr Adolesc Med. 2003 Nov;157(11):1084-8. doi: 10.1001/archpedi.157.11.1084. PMID 14609899
- [Background] Johnston CC, Filion F, Snider L, Majnemer A, Limperopoulos C, Walker CD, Veilleux A, Pelausa E, Cake H, Stone S, Sherrard A, Boyer K. Routine sucrose analgesia during the first week of life in neonates younger than 31 weeks' postconceptional age. Pediatrics. 2002 Sep;110(3):523-8. doi: 10.1542/peds.110.3.523. PMID 12205254
- [Background] Stevens B, Yamada J, Ohlsson A. Sucrose for analgesia in newborn infants undergoing painful procedures. Cochrane Database Syst Rev. 2010 Jan 20;(1):CD001069. doi: 10.1002/14651858.CD001069.pub3. PMID 20091512
- [Derived] Vinall J, Noel M, Disher T, Caddell K, Campbell-Yeo M. Memories of Infant Pain in the Neonatal Intensive Care Unit Influence Posttraumatic Stress Symptoms in Mothers of Infants Born Preterm. Clin J Pain. 2018 Oct;34(10):936-943. doi: 10.1097/AJP.0000000000000620. PMID 29698249
- [Derived] Campbell-Yeo M, Johnston C, Benoit B, Latimer M, Vincer M, Walker CD, Streiner D, Inglis D, Caddell K. Trial of repeated analgesia with Kangaroo Mother Care (TRAKC Trial). BMC Pediatr. 2013 Nov 9;13:182. doi: 10.1186/1471-2431-13-182. PMID 24284002